CLINICAL TRIAL: NCT02238834
Title: A Randomized, Double-blind, Placebo Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of FP-025, an MMP-12 Inhibitor, in Healthy Male Subjects
Brief Title: Phase 1 Safety, Tolerability and Pharmacokinetics (PK) Study of FP-025 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS-Qualitix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP02C-14-001
Record Dates: First submitted 2014-09-05; First posted 2014-09-12 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Phase I; Safety and tolerability; Pharmacokinetic; Randomized; Double Blind; Placebo-Controlled; Single- & Multiple Dose Escalation; FP-025; MMP-12 inhibitor
MeSH Terms: interventions — FP-025

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1-8 Experimental Arm (Experimental)
  Interventions: Drug: FP-025
- SAD Cohorts 1-8 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohorts 1 through 4 Experimental Arm (Experimental): Note: The planned MAD portion of the study was not conducted. Evaluation of FP-025 MAD is being conducted under a separate protocol (Study No. FP02C-17-001).
  Interventions: Drug: FP-025
- MAD Cohorts 1 through 4 Placebo Arm (Placebo Comparator): Note: The planned MAD portion of the study was not conducted. Evaluation of FP-025 MAD is being conducted under a separate protocol (Study No. FP02C-17-001).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FP-025 — Subjects will receive single doses of 200 to up to 800 mg of FP-025 (API-in-capsule) in a dose escalation format (cohorts 1-3). Subjects will receive single doses of 50 to up to 450 mg of FP-025 (ASD-in-capsule) in a dose escalation format (cohorts 4-8).
  Arms: SAD Cohorts 1-8 Experimental Arm
Drug: Placebo — Subjects will receive single doses of FP-025 matching placebo (capsule) in a dose escalation format.
  Arms: SAD Cohorts 1-8 Placebo Arm
Drug: FP-025 — Subjects will receive doses of FP-025 (capsule) twice daily for 5 days.
  Arms: MAD Cohorts 1 through 4 Experimental Arm
Drug: Placebo — Subjects will receive FP-025 matching placebo (capsule) twice daily for 5 days
  Arms: MAD Cohorts 1 through 4 Placebo Arm

SUMMARY:
This is a randomized, placebo controlled, single and multiple ascending dose study to assess the safety and tolerability and pharmacokinetics of FP-025 in healthy subjects.

Note: Dosing in the SAD phase was completed, and the planned MAD portion of the study was not conducted. Evaluation of FP-025 MAD is being conducted under a separate protocol (Study No. FP02C-17-001).

DETAILED DESCRIPTION:
In the SAD part of the study the investigational drug will be administered once in a dose escalation manner starting from 200 mg in Cohort 1 to 2000 mg in Cohort 6. The study drug will be orally taken as capsules. In the MAD part of the study the investigational drug will be administrated twice daily for 5 days depending on the half-life of FP-025, as determined in the SAD part of the study. Study subjects will be randomized in a 1:3 ratio to either placebo or FP-025 in every cohort of the SAD and MAD part of the study.

Note: Dosing in the SAD phase was completed, and the planned MAD portion of the study was not conducted. Evaluation of FP-025 MAD is being conducted under a separate protocol (Study No. FP02C-17-001).

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥20 and ≤65 years with a BMI ≥18 kg/m2 and ≤30 kg/m2.
* A resting pulse ≥50 bpm and ≤100 bpm at the Screening Visit.
* A resting systolic blood pressure of ≤140 mmHg and a resting diastolic blood pressure of ≤90 mmHg at the Screening Visit and the Safety Baseline Visit.
* Baseline laboratory test values within reference ranges based on the blood and urine samples taken at the Screening Visit. Out of normal ranges values (except for liver parameters) may be accepted by the investigator, if not clinically significant.
* The subject is, in the opinion of the investigator, generally healthy based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
* Adequate contraception (double-barrier) will be applied during and until 3 months after completion of the study.
* Signed Informed Consent prior to any study related procedures.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* The subject has taken prescription or non-prescription medication, herbal remedies, vitamins or minerals within 2 weeks prior to the first dose of study product (or within 5 half-lives prior to inclusion for any medication ingested, whichever is longer).
* The subject has a substance abuse-related disorder or has a significant history of drug or alcohol abuse, or a history of drug abuse or a history of substance abuse deemed significant by the investigator.
* The subject should avoid alcohol for at least 5 days before admission into the clinic.
* The subject has taken any investigational products within 30 days prior to the first dose of study product.
* The subject has a history of severe drug allergy or hypersensitivity or food allergy.
* The subject has a history or presence of any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (in particular diabetes or pre-diabetes), haematological, dermatological, venereal, neurological, chronic infectious or psychiatric disease or other major disorder.
* The subject has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, which has not been in remission for at least 5 years prior to the first dose of study product.
* The subject has a history of abdominal surgery (excluding laparoscopic cholecystectomy or uncomplicated appendectomy) or thoracic or non-peripheral vascular surgery within 6 months prior to the first dose of study product.
* The subject has any concurrent illness that may affect the particular target or absorption, distribution, and elimination of the study product.
* The subject has had a clinically significant illness within 4 weeks prior to the first dose of study product.
* The subject has had surgery or trauma with significant blood loss within the last 3 months prior to the first dose of study product.
* The subject has donated blood more than 250 mL within 2 months prior to the first dose of study product.
* The subject has tested positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV).
* The subject is a current smoker or uses other nicotine containing products. Ex-smokers must have ceased smoking at least 6 months prior to the first dose of study product (+ <10 pack years).
* The subject has tested positive at the Screening Visit and at the Safety Baseline Visit for drugs of abuse (amphetamine, cannabinoid, cocaine, morphine, and phencyclidine).
* The subject's corrected QT interval (QTc) (Bazett's or Fridericia's correction) is >450 ms as read on the printout of the ECG produced by the ECG equipment and evaluated by the investigator at the Screening Visit and at the Safety Baseline Visit. An out-of-range or abnormal ECG may be repeated. In total, 3 ECGs should be recorded consecutively and the investigator must evaluate the triplicate ECG. If the subject's QTc is >450 ms on at least 2 ECGs, the subject must be excluded.
* The subject exercises extensively (e.g. marathon, triathlon or other similar high energetic sports). In general, subjects should refrain from sporting for at least 4 days before participation to the study.
* The subject is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.
* A history of psychiatric diseases, i.e depression and/or anxiety related illness.
* Serum creatinine, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above the upper limit of normal (ULN) and deemed clinically significant by the investigator at screening and at the Safety Baseline Visit.
* Hemoglobin, white blood cells (WBC) or platelet count below the lower limit of normal (LLN) and deemed clinically significant by the investigator at screening and at the Safety Baseline Visit.
* Other laboratory results which are clinically significant abnormal at screening and at the Safety Baseline Visit.
* Legal incapacity or limited legal capacity at screening and at the Safety Baseline Visit.
* Employees of the investigator or study centre, as well as first grade family members of the employees or the investigator.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Single ascending dose (SAD): Safety and tolerability of FP-025 | 9 days
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs, and ECG monitoring
Multiple ascending dose (MAD): Safety and tolerability of FP-025 | 13 days
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs, and ECG monitoring

SECONDARY OUTCOMES:
Single ascending dose (SAD): Pharmacokinetics of FP-025 | 2 days
  Plasma concentrations of FP-025
Multiple ascending dose (MAD): Pharmacokinetics of FP-025 | 6 days
  Plasma concentrations of FP-025

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Abd-Elaziz K, Voors-Pette C, Wang KL, Pan S, Lee Y, Mao J, Li Y, Chien B, Lau D, Diamant Z. First-in-Man Safety, Tolerability, and Pharmacokinetics of a Novel and Highly Selective Inhibitor of Matrix Metalloproteinase-12, FP-025: Results from Two Randomized Studies in Healthy Subjects. Clin Drug Investig. 2021 Jan;41(1):65-76. doi: 10.1007/s40261-020-00981-9. Epub 2020 Dec 17. PMID 33331980